CLINICAL TRIAL: NCT02228005
Title: The Effect of a Selective Serotonin Reuptake Inhibitor on Gait, Balance, and Bone Metabolism in Older Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DF-2013-10
Record Dates: First submitted 2014-07-23; First posted 2014-08-28 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2015-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Depression (Experimental): Sertraline 50- 200mg
  Interventions: Drug: Sertraline
- Comparison group (non-depressed) (No Intervention): No intervention

INTERVENTIONS:
Drug: Sertraline — Protocolized titration from 50 to max 200mg based on response and tolerance.
  Other Names: Zoloft
  Arms: Depression

SUMMARY:
The purpose of this study is to examine the effects of sertraline treatment of depression in older adults on gait stability, balance recovery reactions, and markers of bone metabolism. This is a pilot study that will determine feasibility and generate hypotheses for a larger definitive study.

DETAILED DESCRIPTION:
Selective serotonin reuptake inhibitors (SSRIs) are a class of antidepressant medication frequently used to treat depressive and anxiety disorders in the elderly. Although widely considered to be a safe option, several observational studies have found that SSRIs have as strong an association with falls as other psychotropic medications including tricyclic antidepressants and benzodiazepines. However, the potential mechanism for a link between SSRIs and falls is unclear. Compared to other psychotropic medications, SSRIs have lower rates of side effects that could contribute to falls, including sedation, orthostatic blood pressure changes, and anticholinergicity. Interestingly, SSRIs have also been associated with fractures, more so than other classes of antidepressants, in both administrative database studies and prospective cohort studies that control for falls history. Serotonin is known to play a role in regulating bone mass and some studies have found a loss of bone mass in individuals on SSRI treatment.

The association of SSRIs with falls and fractures is confounded by depression which is itself associated with falls, gait instability, bone loss and fractures. The goal of this study is to disentangle the contribution of the disease versus the treatment to risk of falls and fractures. As a first step towards this goal, this pilot study will: i) estimate effect sizes for statistical power calculations for an adequately powered study; and ii) examine the feasibility of timely recruitment of older patients with major depression who have not taken antidepressant medication for a minimum of 2 weeks prior to entering the study.

To address our research question, we have designed a prospective observational pilot study. Older adults with depression will be assessed at baseline, and then 3,6, and 12 weeks after initiation of sertraline antidepressant therapy. A non-depressed comparison group will be used to control for the learning effects of repeated assessment. The outcomes of interest are changes in gait, static balance, and dynamic balance recovery reactions. Our primary outcomes are the short-term changes in these variables at 3 weeks, but we will also perform a longitudinal analysis to assess change over 12 weeks.

ELIGIBILITY:
Depressed group

Inclusion Criteria:

* Clinical diagnosis of Major Depression
* English-speaking
* If currently on an antidepressant, willing to undergo a 2 week washout.

Exclusion Criteria:

* Lifetime bipolar disorder
* Current psychotic disorder or substance use disorder
* Dementia
* Poor baseline mobility or baseline severe gait disorder
* On treatment with fluoxetine or mood stabilizer
* Severe renal impairment, bleeding disorder, recent gastric bleeding or hemorrhagic stroke in past 3 months
* Poor response or serious adverse event with sertraline in the past.

Comparison group

Inclusion Criteria:

- English-speaking

Exclusion Criteria:

* Lifetime diagnosis of depression or dementia
* Currently on antidepressant medication or mood stabilizer
* Poor baseline mobility or baseline severe gait disorder

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in number of steps to recover balance compared to baseline | Baseline, 3 weeks
  Number of steps

SECONDARY OUTCOMES:
Change in CTX-I (Serum collagen type-I cross-linked C-telopeptide) | 12 weeks
  pg/ml
Change in P1NP (Serum procollagen type-1 N-terminal polypeptide) | 12 weeks
  ng/ml
Change in stride variability from baseline | Baseline, 3 weeks
  ms
Change in centre of pressure sway velocity under dual task conditions | Baseline, 3 weeks
  cm/s

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Iaboni, MD DPhil, Principal Investigator — University Health Network and University of Toronto
Locations (1):
- Toronto Rehabilitation Institute, University Health Network, Toronto, Ontario, Canada